CLINICAL TRIAL: NCT05297877
Title: Use of Artificial Intelligence Cardiac Ultrasound Technology in Teaching Point of Care Cardiac Ultrasound - a Randomised Controlled Trial
Brief Title: Use of Artificial Intelligence Cardiac Ultrasound Technology in Teaching Point of Care Cardiac Ultrasound
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National University of Singapore (Other)
Responsible Party: Principal Investigator, NUS Anaesthesia, Principal Investigator, National University of Singapore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: NUS-IRB-2021-484
Record Dates: First submitted 2022-03-07; First posted 2022-03-28 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Cardiac
Keywords: Cardiac Ultrasound

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AI Machine (Experimental): All study participants will undergo a full day (roughly 8 hours) training programme consisting of a pre-test MCQ, a didactic lecture, hands-on training session, a post-test MCQ, and a practical evaluation. They will be randomised to using an A.I. ultrasound machine for teaching.
  Interventions: Other: Experimental AI Echo Machine
- Conventional Machine (Other): All study participants will undergo a full day (roughly 8 hours) training programme consisting of a pre-test MCQ, a didactic lecture, hands-on training session, a post-test MCQ, and a practical evaluation. They will be randomised to using a conventional ultrasound machine for teaching.
  Interventions: Other: Conventional Echo Machine

INTERVENTIONS:
Other: Experimental AI Echo Machine — Participants will go through the training programme using an AI machine for learning.
  Arms: AI Machine
Other: Conventional Echo Machine — Participants will go through the training programme using a conventional machine for learning.
  Arms: Conventional Machine

SUMMARY:
The aim of the study is to evaluate the effectiveness of artificial intelligence (A.I.) cardiac ultrasound technology in teaching point of care cardiac ultrasound (POCUS Cardiac).

ELIGIBILITY:
Inclusion Criteria:

* Medical students with no prior training in point of care cardiac ultrasound

Exclusion Criteria:

* Medical students who have received prior training in point of care cardiac ultrasound
* Participants who are unable to complete the entire training programme (pre-training MCQ, simulation session, post-training MCQ, practical evaluation, follow up practical evaluation one month later)

Ages: 19 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-01-14 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of artificial intelligence (A.I.) cardiac ultrasound technology in teaching point of care cardiac ultrasound vs conventional echo machine | Study till 1 month post-study
  Evaluate the effectiveness between AI and conventional echo machine by pre and post-session MCQs, and post intervention evaluation of practical skills using echo machine

CONTACTS AND LOCATIONS:
Overall Officials: Suresh Paranjothy, Principal Investigator — National University Health System
Locations (1):
- National University of Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No